CLINICAL TRIAL: NCT00346697
Title: A Randomized, Double-Blind, Placebo-Controlled Study of N-3 Fatty Acid on Plasma Triglyceride Levels in Hypertriglyceridemic HIV Patients Receiving Highly Active Antiretroviral Therapy
Brief Title: Omega-3 Fatty Acids for High Triglycerides in HIV-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brown, Todd, M.D., Ph.D. (Individual)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Todd T. Brown, MD, PhD, Associate Professor of Medicine and Epidemiology, Brown, Todd, M.D., Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23AT002862-01 (NIH); K23AT002862-01 (NIH)
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: HIV Infections; AIDS; Dyslipidemia; Hypertriglyceridemia
Keywords: AIDS; HIV; HAART; Lipids; Triglycerides; Cholesterol; omega-3 fatty acids; bone turnover; inflammation; insulin resistance
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Dyslipidemias; Hypertriglyceridemia; Inflammation; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LOVAZA (Experimental): 4 g/d of omega-3 fatty acid esters, plus dietary counseling
  Interventions: Drug: Omega-3 fatty acid administration
- Placebo (Placebo Comparator): Corn oil placebo, plus dietary counselling
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 fatty acid administration — LOVAZA 1 gram capsules, 4 capsules daily
  Arms: LOVAZA
Drug: Placebo — Corn-oil placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of omega-3-fatty acids in HIV-infected patients with hypertriglyceridemia. In addition, we, the researchers, will evaluate the effect of omega-3 fatty acid administration of markers of bone turnover and inflammation.

DETAILED DESCRIPTION:
Hypertriglyceridemia is common among HIV-infected patients receiving Highly Active Antiretroviral Therapy (HAART). Although fibrates, statins, and niacin have all been used in the management of hypertriglyceridemia in HIV-infected patients, optimal control is difficult to achieve and other agents are needed. Omega-3 fatty acids are effective for lowering triglycerides in patients without HIV infection, but experience in HIV-infected patients is limited. In addition, omega-3 fatty acids may also have secondary benefits in decreasing bone resorption and decreasing markers of systemic inflammation. The purpose of this study is to evaluate the efficacy and safety of omega-3-fatty acids in HIV-infected patients with hypertriglyceridemia. In addition, we will evaluate the effect of omega-3 fatty acid administration of markers of bone turnover and inflammation. It is 8- week randomized, double-blind trial of omega-3 fatty acids (LOVAZA, GSK, Inc) compared to placebo in 48 HAART-treated HIV-infected patients with triglycerides between 250 and 1000 mg/dl receiving dietary counseling. Subjects will be recruited from three centers (Johns Hopkins, Georgetown, and Los Angeles VAMC). The primary endpoint will be the change in triglyceride concentrations from baseline in the LOVAZA group compared to the placebo group. Secondary endpoints include the effect of LOVAZA on other lipid targets (total cholesterol, LDL cholesterol, HDL-cholesterol), markers of systemic inflammation, markers of bone turnover, markers of insulin resistance, HIV-disease control (CD4+ counts, HIV viral loads), measures of hepatotoxicity (ALT), platelet function, and patient reports of adverse events. Omega-3 fatty acids may be a useful adjunct in the treatment of hypertriglyceridemia in HIV-infected patients, but additional controlled studies are needed to assess its safety and efficacy using a purified, standardized preparation.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give informed consent
* Age ≥ 18 years
* HIV-1 infection documented at any time prior to study entry
* Fasting plasma triglyceride value between 200 and 1000 mg/dL on two occasions within 4 weeks
* Subjects must be receiving a stable antiretroviral medication regimen for > 3 months without any anticipated changes during the study interval
* Females must not be pregnant or lactating. Females of childbearing potential and males must use a reliable means of contraception
* On stable lipid modification pharmacotherapy for at least 8 weeks prior to study entry

Exclusion Criteria

* Hemoglobin A1C > 8.5 %
* Uncontrolled hypothyroidism (TSH > 4.5)
* HIV viral load > 5,000 copies/ml (cpm),
* Active liver disease and/or liver transaminases greater than 2.0 X upper limit of normal
* Active kidney disease or serum creatinine > 2.5 mg/dL
* Myocardial infarction, unstable ischemic heart disease, stroke, or coronary revascularization procedure
* Uncontrolled hypertension within 4 weeks of study entry (SBP > 180 mmHg or DBP > 100 mmHg)
* Use of systemic cancer chemotherapy within 8 weeks of study entry
* Pregnancy or breastfeeding
* Drug or alcohol dependence, or other conditions which may affect study compliance
* History of coagulopathy or use of anticoagulants such as warfarin
* Use of omega-3 fatty acid preparation in the 12 weeks prior to randomization
* Significant changes in clinical status from the Screening Visit which would preclude the patient from being an appropriate candidate.
* Any of the following laboratory parameters: hematocrit < 25%, absolute neutrophil count < 1.5 x 10^9/L, platelets < 100 x 10^9/L or hemoglobin < 8.0 gm/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd T. Brown, MD, Principal Investigator — Johns Hopkins University; David Leaf, MD, Principal Investigator — Veterans Adminstration of Greater Los Angeles Health System; Mattew Goetz, MD, Principal Investigator — Veterans Adminstration of Greater Los Angeles Health System; Adrian S Dobs, MD, Principal Investigator — Johns Hopkins University; Joseph Timpone, MD, Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - Veterans Administration of Greater Los Angeles Health System, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Result] Metkus TS, Timpone J, Leaf D, Bidwell Goetz M, Harris WS, Brown TT. Omega-3 fatty acid therapy reduces triglycerides and interleukin-6 in hypertriglyeridemic HIV patients. HIV Med. 2013 Oct;14(9):530-9. doi: 10.1111/hiv.12046. Epub 2013 May 19. PMID 23683266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took plave between November 2006 and September 2010 at 3 sites (Johns Hopkins University, Baltimore, MD;Veteran's Administration Greater Los Angeles Healthcare System (Los Angeles, CA), and the Georgetown University Hospital (Washington, DC). Participants were recruited from the HIV Clinics at these institutions.
Period: Overall Study
Arm/Group | LOVAZA | Placebo
Started | 24 | 24
Completed | 24 | 23
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LOVAZA | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (5.2) | 48.2 (8.0) | 49.2 (6.8)
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [47 to 52] | 48 [41 to 52] | 49.5 [45.5 to 52.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Triglyceride Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 24 | 23
mg/dl | -34 [-149 to 9.5] | 40 [-51 to 123]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Total Cholesterol Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Groups:
- Placebo: Corn oil placebo, plus dietary counselling
  Omega-3 fatty acid administration: LOVAZA 1 gram capsules, 4 capsules daily
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 24 | 23
mg/dl | -16 [-31 to 23] | -5 [-25 to 19]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = .80, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Non-HDL Cholesterol Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 24 | 23
mg/dl | -12.5 [-30 to 17] | -9 [-23 to 21]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in HDL Cholesterol Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 24 | 23
mg/dl | 1.5 [-2 to 4] | -1 [-6 to 3]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in HOMA-IR From Baseline in the LOVAZA Group Compared to the Placebo Group
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
units on a scale | 0.56 [-0.51 to 3.6] | 0.94 [-1.9 to 4.0]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in CD4+ T-cell Counts From Baseline in the LOVAZA Group Compared to the Placebo Group
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: cells/cc
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 21 | 21
cells/cc | 20 [-28 to 107] | 7 [-42 to 118]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in hsCRP Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
ng/ml | -0.04 [-1.19 to 0.35] | 0.17 [-0.38 to 0.99]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in IL-6 Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
pg/mL | -0.62 [-1.89 to 0.13] | 0.19 [-0.13 to 1.65]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in TNF-a Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
pg/mL | -0.36 [-2.27 to 0.014] | 0.58 [-1.15 to 2.25]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in sTNFR1 Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
pg/mL | -0.90 [-91.8 to 69.8] | -66.3 [-189 to 152]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in sTNFR2 Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
pg/mL | -63.5 [-371 to 615] | 118 [-499 to 565]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in CTX Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
ng/mL | -0.02 [-0.08 to 0.02] | 0.03 [-0.06 to 0.09]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change in P1NP Concentrations From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 23 | 22
mcg/L | -5.23 [-12.6 to -0.16] | -2.12 [-8.7 to 1.3]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change in Collagen ADP From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 18 | 16
seconds | 6.5 [-3 to 21] | -6 [-13 to 9.5]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.12, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change in Collagen Epinephrine From Baseline in the LOVAZA Group Compared to the Placebo Group.
Time Frame: 8 weeks
Population: Analysis done on all participants with available data
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | LOVAZA | Placebo
Number analyzed (Participants) | 18 | 16
seconds | 5.5 [-6 to 39] | -18 [-46.5 to 28]
Statistical Analysis 1: Comparison: LOVAZA vs Placebo; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | LOVAZA | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LOVAZA (N=24) | Placebo (N=24)
Gastrointesitnal Side effects (dyspepsia, bloating, fishy taste) (Gastrointestinal disorders) | 3 (3) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No